CLINICAL TRIAL: NCT06291233
Title: A Hybrid Effectiveness-Implementation RCT of Virtual Interview Training for Autistic Transition-Age Youth
Brief Title: Interview TIME: Training Inspired Minds for Employment
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Matthew Smith, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HUM00236812; 1R01MH132656-01 (NIH)
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-02

CONDITIONS: Autism Spectrum Disorder
Keywords: Job interview skills; Students
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Interview Training (Experimental)
  Interventions: Behavioral: Virtual Interview Training (VIT)
- Services-as-usual (Active Comparator)
  Interventions: Behavioral: Services-as-usual

INTERVENTIONS:
Behavioral: Virtual Interview Training (VIT) — Teachers will administer the intervention (Virtual Interview Training) with the student participants. University of Michigan research staff will train all teachers (including sites in California) and will provide support as necessary throughout the intervention delivery process. Surveys will be captures several times throughout delivery as delivery is expected to be anywhere between 4 to 6 weeks long.
  Arms: Virtual Interview Training
Behavioral: Services-as-usual — Participants will receive services-as-usual at participants school or program for approximately 6 weeks. Those that are in the active control group will receive access to the e-learning content of the Rita/Travis intervention (not the practice interviews) and will be able to review the e-learning content with teacher's supervision. In addition, this group will review a series of video conversations with autistic adults about navigating the pathway to a career. Surveys will be collected at different time points after randomization.
  Arms: Services-as-usual

SUMMARY:
The purpose of the study is to see if an internet job interview training program can help people that have autism improve interview skills and access to jobs.

Participants will be randomized to use Virtual Interview Training (VIT) or continue services as usual (active control group).

DETAILED DESCRIPTION:
Participants will have assessments that will be done over the computer or in-person at school or program site. Assessments will be about participants background, employment history, mood and feelings, autistic traits, memory, mental health issues, such as depression and anxiety, and other things. Some assessments will be audio and/or video recorded.

Please note that there will be teachers and staff consented (approximately n=32) to deliver the intervention, however, will not count for the clinical trial. Therefore, the information will not be added to the anticipated enrollment numbers in study design.

ELIGIBILITY:
Inclusion Criteria:

* Participants have a diagnosis on the autism spectrum
* Participants are enrolled in pre-employment transition services
* Participants have at least a third-grade reading level
* Are unemployed or employed and job-seeking

Exclusion Criteria:

- Not enrolled in pre-employment transition services

Ages: 16 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Competitive Employment based on self-report employment surveys | Approximately 9 months after randomization
  Self-report employment surveys completed. Employment will be tracked as 0 (no job) and 1 (job). Higher scores indicate a better outcome.
Change in Job Interview Skills from Mock Interview Rating Scale (MIRS) | Pre-Test (baseline), post-test (approximately 6 weeks)
  Interviewing skills will be measured using a role-play measure in which subjects act out two job interview scenarios with trained actors. Interviews will be video recorded and scored. There is one pre-test score and one post-test score. There are 15 questions on a scale from 1 to 7 (scores range from 15 to 105), with higher scores indicating a better outcome (better interview skills).
Time to Employment | Approximately 9 months after randomization
  The number of days between randomization and obtaining employment using a questionnaire.

SECONDARY OUTCOMES:
Change in Interview Anxiety using a modified version of the brief Personal Report of Public Speaking Apprehension (PRSPA) | Pre-Test (baseline), post-test (approximately 6 weeks)
  This is a 13 item self-report using a modified version of the brief Personal Report of Public Speaking Apprehension (PRSPA). After reviewing the brief PRSPA, the study team selected and reframed 13 items using a three-point Likert-type scale (0 = "not at all," 1 = "sometimes," and 2 = "often"). Higher scores indicated higher anxiety, and scores could range from 0 to 26.
Change in Interview Motivation | Pre-Test (baseline), post-test (approximately 6 weeks)
  This is a 10 item self-report using a five-point Likert scale (1 = Not at all true, 5 = Very true). Higher scores indicate higher job interview motivation, a better outcome, and scores range from 10 to 50)
Change in Work Readiness using the Work Readiness Scale (WRS) | Pre-Test (baseline), post-test (approximately 6 weeks)
  Change in work readiness using the Work Readiness Scale (WRS) which is a 13 item self-report using a five-point Likert scale (1 = Strongly Disagree to 5 = Strongly Agree) with higher scores indicating a higher readiness to work, a positive outcome. Scores range from 13 to 65.
Change in Work Motivation using the Work Motivation Scale (WMS) | Pre-Test (baseline), post-test (approximately 6 weeks)
  Change in work motivation using the Work Motivation Scale (WMS) which is a 12-item self-report using a four-point Likert scale (1 = Disagree to 4 = Strongly Agree) with higher scores indicating a higher motivation to work, a better outcome. Scores range from 13 to 52.
Change in Social Cognition using the Bell-Lysaker Emotion Recognition Task Adult (BLERT-A) | Pre-Test (baseline), post-test (approximately 6 weeks)
  Change in social cognition using the Bell-Lysaker Emotion Recognition Task Adult (BLERT-A). There are 21 videos shown to participants and are scored as either correct (1) or incorrect (0). A total score is provided and can range from 0 to 21, with higher scores indicating a higher social cognition ability, a better outcome.
Change in Interview Knowledge | Pre-Test (baseline), post-test (approximately 6 weeks)
  Change in interview knowledge by using a 10-item survey designed to assess basic knowledge about job interviews. There are multiple choice questions, and answers are marked as either correct (1) or incorrect (0). Higher scores indicate better interview knowledge, a positive outcome. Scores range from 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Smith, Principal Investigator — University of Michigan
Locations (15):
- United States (15):
  - Classical Academy, Oceanside, California
  - Outside the Lens, San Diego, California
  - Transition Resources for Adult Community Education, San Diego, California
  - The Institute for Effective Education, San Diego, California
  - The San Diego State University, San Diego, California
  - Mount Miguel High School, Spring Valley, California
  - Urban Autism Solutions, Chicago, Illinois
  - Ann Arbor Academy, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - Milford High School, Highland, Michigan
  - Lincoln Park, Lincoln Park, Michigan
  - Lakeland High School, White Lake, Michigan
  - Kessler Foundation, East Hanover, New Jersey
  - Banyan High School, Little Falls, New Jersey
  - Alpine Learning Group, Paramus, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
Survey data from the randomized control trial (RCT) participants will be deposited into the National Institute of Mental Health (NIMH) Data Archive repository. This will include basic demographic information and self reported data from validated measures that can be found within the NIMH Data Archive Repository's data dictionaries. Identifiable information will not be available for access.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be made available within 6 months of the study's conclusion and will remain available for at least 5 years.
Access Criteria: According to the NIMH Data Archive Repository, researchers who want to access the data may create a username and password and submit a Data Access Request for permission to access the data. Please see the following website for more details: https://nda.nih.gov/nda/access-data-info